CLINICAL TRIAL: NCT04389502
Title: Efficacy of a Mobile Clinical Decision Support System (CaPtyVa CCR App) to Improve Performance of Gastroenterology and Coloproctology Specialists in Colorectal Cancer Screening and Surveillance According to Guideline Recommendations: A Randomized Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Aleman (Other)
Responsible Party: Principal Investigator, Lisandro Pereyra, MD, Hospital Aleman
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CaPtyVa CCR app
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaPtyVa app group (Experimental): Those assigned to the CaPtyVa app group will receive a tutorial video describing its operation and will have to complete 10-item clinical vignette quiz according to the app recommendations based on local current CRC screening and surveillance guidelines on every question. Physicians in this group will download a free of charge application (CaPtyVa CCR APP, Digital Means, Argentina) on their iOs or Android device.
  Interventions: Device: CaPtyVa app
- Control group (Active Comparator): The ones assigned to the control group will be asked to complete the 10-item clinical vignette quiz according to their current knowledge on local current CRC screening and surveillance guidelines
  Interventions: Other: Control group

INTERVENTIONS:
Device: CaPtyVa app — The apps stores all the current local Clinical practice guidelines information related to CRC screening and surveillance and through its decision algorithms assist physicians in the screening process. In the screening function, CaPtyVa helps the physicians to classify patient´s according to their individual CRC risk and to determine how and when to start with screening tests. In the surveillance, function the app assist the physician in determining when to repeat the next colonoscopy according to guideline recommendation
  Arms: CaPtyVa app group
Other: Control group — current physician knowledge on local current CRC screening and surveillance guidelines
  Arms: Control group

SUMMARY:
This prospective study evaluates the use of a (Mobile Decision Support Systems), MDSS (CaPtyVa CCR app) in order to improves gastroenterology and coloproctology specialist's performance in CRC screening and surveillance according to local current guidelines.

DETAILED DESCRIPTION:
The proper implementation of clinical practice guidelines (CPGs) has the potential to improve health care quality and reduce costs by promoting the use of evidence-based interventions. However, these benefits vary largely according to the way CPGs are put into effect. The behavior of physicians towards CPGs is a determining factor in their successful implementation. It has been suggested that physicians have difficulties in memorizing and processing the complex information contained in CPGs.

Computer-Based Clinical Decision Support Systems (CDSSs) are defined as "any software designed to aid in clinical decision making in which characteristics of individual patients are matched to a computerized knowledge. These systems have shown to: improve prescribing practices, reduce serious medication errors, enhance the delivery of preventive care services, and improve adherence to recommended care standards.

Recent evidence had also suggests that mobile technologies could provide an effective approach in order to allow these Decision Support Systems to be implemented (Mobile Decision Support Systems, MDSS) without requiring personal computers or its integration into other clinical information systems.

Colorectal cancer (CRC) is a global major medical and public health challenge, accounting for 881.000 deaths annually. Evidence-based CRC screening strategies have shown to be effective in reducing CRC mortality. Hence, the majority of CRC deaths are believed to be the result of CRC screening process breakdowns. Multiple studies report overuse and underuse of colonoscopy, as well as poor physician's knowledge about CRC screening CPG's and their inability to apply them in daily clinical practice. All these factors may threaten the effectiveness of CRC screening programs.

The above mentioned problematic added to recent evidence showing a strong willingness of the physicians to use mobile-based apps in order to assist them in making guideline-concordant recommendations, motivated us to satisfy this need and we developed the first MDSS(CaPtyVa CCR app), to assist physicians in the CRC screening and surveillance task process.

The aim of this prospective study is to evaluate whether a MDSS (CaPtyVa CCR app) improves gastroenterology and coloproctology specialist's performance in CRC screening and surveillance according to local current guidelines

A prospective, nationwide, single blinded, randomized study will be conducted. A 10-question anonymous survey was created with CRC screening and surveillance clinical vignettes reflecting real life daily practice scenarios. After the question were developed, they were pre-tested and discussed for content and clarity by three experienced gastroenterologists. Gastroenterologists and coloproctologists; randomly selected will be invited by e-mail to participate in this study between May 2020 and June 2020.

ELIGIBILITY:
Inclusion Criteria:

* Gastroenterologists and coloproctologists members of four medical societies from Argentina and Uruguay: Endoscopistas de Buenos Aires(ENDIBA), Federación Argentina de Endoscopía Digestiva(FAED), Sociedad Argentina de Coloproctología(SACP) and Sociedad Uruguaya de Endoscopía Digestiva(SUED)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Correct Answers (60% group) | 1 month
  Proportion of physicians correctly answering at least 60% of the clinical vignettes according to local current guidelines. Responses consistent with the current CRC screening and surveillance guidelines of the Instituto Nacional del Cancer (INC) of Argentina are considered accurate

SECONDARY OUTCOMES:
Correct Answers (80% group) | 1 month
  Proportion of physicians correctly answering at least 80% of the clinical vignettes according to the guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Aleman, CABA, Argentina

IPD SHARING:
Plan to Share IPD: No